CLINICAL TRIAL: NCT03051308
Title: University of Wisconsin Solution Versus New Parathyroid Transport Solution for Parathyroid Allotransplantation: Effects on Calcium Sensing and Vitamin D Receptor During Cold Ischemia
Brief Title: University of Wisconsin Solution Versus New Parathyroid Transport Solution for Parathyroid Allotransplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SB Istanbul Education and Research Hospital (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Erhan Aysan, Principal Investigator, SB Istanbul Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BAVUvsUW
Record Dates: First submitted 2017-01-29; First posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Parathyroid Allotransplantation
Keywords: Parathyroid cell viability; Ischemia; Parathyroid allotransplantation; Vitamin D Receptor; Calcium Sensing Receptor
MeSH Terms: conditions — Ischemia | interventions — University of Wisconsin-lactobionate solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- First Application in Hour 0 (Experimental): Viability, Calcium-sensing receptor, Vitamin D receptor and parathormone levels of Parathyroid cells (10^7 cells) at 'First Application in Hour 0' non-cold ischemia tissue group
  Interventions: Combination Product: NPT and UW Solution
- First Application in Hour 6 (Experimental): Viability, Calcium-sensing receptor, Vitamin D receptor and parathormone levels of Parathyroid cells (10^7 cells) at 'First Application in Hour 6' cold ischemic tissue group
  Interventions: Combination Product: NPT and UW Solution
- First Application in Hour 12 (Experimental): Viability, Calcium-sensing receptor, Vitamin D receptor and parathormone levels of Parathyroid cells (10^7 cells) at 'First Application in Hour 12' cold ischemic tissue group
  Interventions: Combination Product: NPT and UW Solution
- First Application in Hour 18 (Experimental): Viability, Calcium-sensing receptor, Vitamin D receptor and parathormone levels of Parathyroid cells (10^7 cells) at 'First Application in Hour 18' cold ischemic tissue group
  Interventions: Combination Product: NPT and UW Solution
- First Application in Hour 24 (Experimental): Viability, Calcium-sensing receptor, Vitamin D receptor and parathormone levels of Parathyroid cells (10^7 cells) at 'First Application in Hour' 24 cold ischemic tissue group
  Interventions: Combination Product: NPT and UW Solution

INTERVENTIONS:
Combination Product: NPT and UW Solution — Tissue preservation solutions for transplantation

SUMMARY:
Compare the functionality of new parathyroid transport solution (NPTS) with University of Wisconsin Solution (UW) on parathyroid glands. Also assess its effects on cell viability, parathormone (PTH) secretion, calcium-sensing receptor (CaSR) and vitamin D receptor (VDR) levels during cold ischemia.

DETAILED DESCRIPTION:
Parathormone (PTH) and vitamin D are two critical hormonal regulators of calcium homeostasis. There is an important relationship between the PTH release and vitamin D receptor for controlling hormonal systems. Also calcium-sensing receptor plays a crucial role in regulating parathormone secretion which means controlling the calcium-dependent systemic ion homeostasis.

Cold ischemia protects organs and tissues by slowing their metabolism. The cold ischemia of the transplant tissue is a very important process. The University of Wisconsin (UW) solution substantially improves graft preservation and consequently increases patient survival. The researchers newly developed NPTS for transportation of parathyroid glands.

For the comparision the researchers measured the parathyroid cell viability and the calcium sensing and vitamin D receptor density of the parathyroid cells at the 0, 6, 12 and 24 hours of cold ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have parathyroid hyperplasia due to chronic renal failure.

Exclusion Criteria:

* Patients who refused to join the study
* Patients younger than 18 years and older than 80 years.
* Patients who have hepatitis B,
* Patients who have hepatitis C,
* Patients who have human immunodeficiency virus (HIV).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2017-06-01 (Estimated); Study Completion 2017-07-01 (Estimated)

PRIMARY OUTCOMES:
Cell viability of Parathyroid cells after isolation process | 0 hour
  After removal of hyperplastic parathyroid glands, each gland will keep in ice cold NPTS and UW solution for transportation to laboratory.
  Then the investigators will measure the viability of Parathyroid cells after isolation process.
Cell viability of Parathyroid cells after 6 hour of cold ischemia | 6 hour
  After removal of hyperplastic parathyroid glands, each gland will keep in ice cold NPTS and UW solution for transportation to laboratory. After 6 hours the investigators will measure the viability of Parathyroid cells after isolation process.
Cell viability of Parathyroid cells after 12 hour of cold ischemia | 12 hour
  After removal of hyperplastic parathyroid glands, each gland will keep in ice cold NPTS and UW solution for transportation to laboratory. After 12 hours the investigators will measure the viability of Parathyroid cells after isolation process.
Cell viability of Parathyroid cells after 18 hour of cold ischemia | 18 hour
  After removal of hyperplastic parathyroid glands, each gland will keep in ice cold NPTS and UW solution for transportation to laboratory. After 18 hours the investigators will measure the viability of Parathyroid cells after isolation process.
Cell viability of Parathyroid cells after 24 hour of cold ischemia | 24 hour
  After removal of hyperplastic parathyroid glands, each gland will keep in ice cold NPTS and UW solution for transportation to laboratory. After 24 hours the investigators will measure the viability of Parathyroid cells after isolation process.

SECONDARY OUTCOMES:
Parathormone Release of Parathyroid Cells | 1 day
  The investigators will measure the parathormone level from cultured parathyroid cells

CONTACTS AND LOCATIONS:
Overall Officials: Erhan Aysan, Prof. M.D., Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Belzer FO, Southard JH. Principles of solid-organ preservation by cold storage. Transplantation. 1988 Apr;45(4):673-6. doi: 10.1097/00007890-198804000-00001. No abstract available. PMID 3282347
- [Background] Southard JH, van Gulik TM, Ametani MS, Vreugdenhil PK, Lindell SL, Pienaar BL, Belzer FO. Important components of the UW solution. Transplantation. 1990 Feb;49(2):251-7. doi: 10.1097/00007890-199002000-00004. PMID 1689516
- [Background] Guibert EE, Petrenko AY, Balaban CL, Somov AY, Rodriguez JV, Fuller BJ. Organ Preservation: Current Concepts and New Strategies for the Next Decade. Transfus Med Hemother. 2011;38(2):125-142. doi: 10.1159/000327033. Epub 2011 Mar 21. PMID 21566713
- [Background] Voigt MR, DeLario GT. Perspectives on abdominal organ preservation solutions: a comparative literature review. Prog Transplant. 2013 Dec;23(4):383-91. doi: 10.7182/pit2013100. PMID 24311404